CLINICAL TRIAL: NCT05382572
Title: Pulmonary Fibrosis Foundation Community Registry
Status: Recruiting | Type: Observational
Sponsor: Pulmonary Fibrosis Foundation (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: HUM00202724
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Fibrosis; Interstitial Lung Disease; Lung Fibrosis; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: An individual diagnosed with PF or ILD, including those who are post lung transplant.
- Family Members: A family member (defined as biological parent, full or half-sibling, or biological child) of an individual with PF or ILD.
- Caregivers: An individual who has cared (currently or in the past) for an individual with PF or ILD.

SUMMARY:
Pulmonary fibrosis (PF) results from a diverse group of health conditions and affects the lives of patients (including those who are post lung transplant), caregivers and family members. The Pulmonary Fibrosis Foundation Community Registry will offer an online portal where participants can self-enroll and directly contribute information about their experience with PF to be compiled into a longitudinal data set for use by researchers.

DETAILED DESCRIPTION:
The PFF Community Registry is an observational, longitudinal cohort study. The Community Registry will enroll three different cohort groups:

1. Patients with PF, including those who are post lung transplant
2. Caregivers of patients with PF
3. Family members of patients with PF

This is an online registry open to individuals affected by PF in the US. It is not associated with a physical location or institution. Individuals may self-enroll online and contribute data to the Community Registry by answering a series of surveys at regular intervals.

Participants may also elect to be contacted about future research projects through the PFF Community Registry portal. However, this is not required to participate in the Community Registry itself.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form online
2. Male or female, aged 18 or older
3. Affected by PF as a member of at least one of the following cohorts:

   1. An individual diagnosed with PF or ILD, including those who are post lung transplant, or
   2. An individual who has cared (currently or in the past) for an individual with PF or ILD, and / or
   3. A family member (defined as parent, full or half-sibling, or child) of an individual with PF or ILD.
4. Has internet access and a valid email address.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Primary residence or place of care is outside of the US.
2. Inability or unwillingness of a participant to provide informed consent or comply with study protocol.
3. Any condition or circumstance not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
4. Patients who were diagnosed with any of the below lung diseases. Similarly caregivers and family members associated with these diseases would be excluded.

   * Sarcoid
   * Lymphangioleiomyomatosis (LAM)
   * Pulmonary alveolar proteinosis (PAP)
   * Cystic fibrosis (CF)
   * Amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Community Registry will enroll three different cohort groups:
  1. Patients with PF or ILD, including those who are post lung transplant
  2. Caregivers of patients with PF or ILD
  3. Family members of patients with PF or ILD
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have or had interstitial lung disease (ILD) enrolled in the PFF Community Registry | 3 years
Number of caregivers of patients who have or had ILD enrolled in the PFF Community Registry | 3 years
Number of family members of patients who have or had ILD enrolled in the PFF Community Registry | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Flaherty, MD, Study Chair — Pulmonary Fibrosis Foundation
Locations (1):
- Pulmonary Fibrosis Foundation, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pulmonary Fibrosis Foundation Registry Information — https://www.pulmonaryfibrosis.org/pff-registry/for-researchers